CLINICAL TRIAL: NCT07337382
Title: The Optimising Isolation, Quarantine and Distancing Study for COVID-19
Acronym: Optimise
Status: Active, not recruiting | Type: Observational
Sponsor: Macfarlane Burnet Institute for Medical Research and Public Health Ltd (Other)
Collaborators: The Peter Doherty Institute for Infection and Immunity (Other); University of Melbourne (Other); Swinburne University of Technology (Other); La Trobe University (Other); Monash University (Other); SNA Toolbox (Unknown); Centre for Culture, Ethnicity & Health (Unknown); Macquarie Group Foundation (Unknown); Victorian State Government (Unknown)
Responsible Party: Sponsor
Other Study IDs: 202006
Record Dates: First submitted 2020-11-05; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-10

CONDITIONS: COVID19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Observational Group 1: Group 1/Seed set 1 - recently diagnosed 'COVID-19 cases' (Group 1) and their social network with up to 2 waves of /Key people, will be followed up for 1 month initially with specific monitoring tools before they will transition into ongoing follow up and monitoring as recruitment group 2
- Observational Group 2: Group 2/Seed set 2 - people from the general community that are not currently infected with COVID19 'Group 2' that are practicing physical distancing and represent specific key risk groups, and their social network with up to 2 waves of Key people

SUMMARY:
The Australian government swift interventions and actions early to the COVID 19 epidemic included enforced quarantine, isolation, varying degrees of social and physical distancing measures, travel restrictions, community level testing and enhanced contact tracing models which effected the trajectory of the epidemic impact. While the search for effective therapeutics and vaccines continues, it is important to understand how to effectively implement and optimise the current public health interventions available; application of traditional contact tracing , contributions of new contact tracing mobile phone applications, community level testing and use of specific fit for purpose diagnostic tests; to screen, detect and provide evidence of infection clearance. While the suppression measures have been effective on disease transmission rates, it has had economic, social and non COVID-19 health costs impacts. As community restrictions change it will be important to monitor and evaluate the effectiveness of these key interventions. This is a longitudinal study that will follow the experience and behaviors of 2 key risk populations impacted by COVID-19 transmission containment measures.

DETAILED DESCRIPTION:
This is a mixed methods longitudinal study of a cohort of 1000 participants for a 12 month period. Victorian adults from three key risk populations will be recruited into two longitudinal cohort groups. It will follow the experiences and behaviors of the groups;

Recruitment group 1/Seed set 1 - recently diagnosed 'COVID-19 cases' (Group 1) and their social network with up to 2 waves of /Key people, will be followed up for 1 month initially with specific monitoring tools before they will transition into ongoing follow up and monitoring as recruitment group 2

Recruitment group 2/Seed set 2 - people from the general community that are not currently infected with COVID19 'Group 2' that are practicing physical distancing and represent specific key risk groups, and their social network with up to 2 waves of Key people.

Oversampling of vulnerable populations including people with disabilities, single parents and people living alone will be conducted across all groups.

Individuals may be invited to participate in more than one cohort when they change between risk population definitions.

The project aims to meet the following objectives using a longitudinal cohort design and a mixed method of qualitative and quantitative tools to enable us to assess changes within individuals over time and to assess the influence of social networks on their health, well-being, attitudes and perceptions. To assess the feasibility, acceptability and implementation of new interventions designed to support a reduction in disease transmission, including testing strategies, we will recruit a small sub-sample of participants into a sub-studies that will assess implementation outcomes.

Objectives of the study are:

1. To assess adherence to government intervention strategies (i.e. early testing, isolation and physical distancing) and identify factors that promote/inhibit compliance to intervention strategies designed to reduce transmission.
2. To better understand, assess and monitor the unintended health, social and economic consequences of the government interventions to control COVID-19 transmission
3. To collect and collate empirical data regarding transmissions dynamics, social contacts and mixing patterns of COVID19 cases , their contacts and key vulnerable groups to develop and refine mathematical models that will improve the precision and timeliness of dynamic transmission estimates
4. To test the acceptability, feasibility and effectiveness of (i) new and existing diagnostic tests and testing strategies and (ii) new and existing intervention strategies (therapeutic, behavioural, social) to support early diagnosis and subsequently reduce transmission.

ELIGIBILITY:
Inclusion Criteria:

Community participants -

Exclusion Criteria:

Unable to provide consent -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants adults living in Victoria
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-09-30 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from response in baseline questionnaires to Adherence (non-adherence) with COVID19 transmission containment measures | 18 months
  Participants will complete behavioural questionnaires and diaries as binary daily measure of outcomes of compliance/non-adherence for each individual, determined by their ability to adhere to government regulations
Change from response in baseline questionnaires depicting what are the unintended health, social and economic consequences of the government response to control COVID19 transmission | 18 months
  Participants will complete behavioural questionnaires and diaries. e.g. Anxiety (using GAD scale: https://patient.info/doctor/generalised-anxiety-disorder-assessment-gad-7).
What are the social contacts and mixing patterns of COVID-19 cases | 18 months
  The behavioural questionnaire participants will be ask to complete include nominating the number of social network contacts per day.
What are the types of social contacts and mixing patterns of COVID-19 cases | 18 months
  The questionnaire participants will be ask to complete will include nominating the relationship with their contacts per day(i.e. partner, child, friend), and individuals COVID test status, providing detailed specifics of the projects social network data.
Measure of the efficacy of government interventions, | 18 months
  Participants responses to behavioural questionnaires and focus group discussions will be used as binary measurers; including but not limited to the number/proportion of participants who receive a score indicating accurate knowledge of government recommendations, receive a score of using COVID-19 prevention measures as recommended by the government.

SECONDARY OUTCOMES:
Collect data of positive COVID19 cases reported in study participant questionnaires. | 18 months
  The COVID 19 data will be analysed to determine the cases reported and if there are social contacts nominated in the questionnaires showing any linkage of cases. The social mixing patterns nominated of COVID19 cases, will be used to develop and refine mathematical models to improve precision and timeliness of dynamic transmission estimates.
Assess the effectiveness of government interventions to reduce COVID-19 transmission from questionnaire responses from cohort participants | 18 months
  Including but not limited to the number/proportion of participants with accurate knowledge of government recommendations and the number/proportion of participants using COVID-19 prevention measures as recommended by the government.
To investigate new and alternative tests to diagnose COVID-19. | 18 months
  Participants of the Optimise main study who are diagnosed with COVID-19 and their contacts will be invited to participate in a sub study of saliva testing compared with deep nasal/throat swab testing for the diagnosis of COVID-19 using RT-PCR

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - The Macfarlane Burnet Institute for Medical Research and Public Health, Melbourne, Victoria
  - The Peter Doherty Institute for infection and immunity, Melbourne, Victoria